CLINICAL TRIAL: NCT01180296
Title: Prevention of Recurrent Preterm Birth With Micronized Progesterone
Brief Title: Oral Progesterone for Prevention of Preterm Birth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fetal Medicine Foundation (Other)
Responsible Party: Principal Investigator, David S. McKenna, PI, Fetal Medicine Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MVH-MP-Pilot-RCT
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Preterm Birth
Keywords: Preterm birth, prevention, progesterone, oral
MeSH Terms: conditions — Premature Birth | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progesterone Group (Experimental): Oral Micronized Progesterone
  Interventions: Drug: oral micronized progesterone
- Placebo (Placebo Comparator): Identical Placebo Tablet
  Interventions: Drug: Identical Placebo tablet

INTERVENTIONS:
Drug: oral micronized progesterone — oral micronized progesterone = 400 mg oral micronized progesterone nightly from 16 to 34 weeks
  Other Names: Prometrium(TM)
  Arms: Progesterone Group
Drug: Identical Placebo tablet — Identical Placebo tablet = placebo taking nightly from 16 to 34 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
To evaluate whether daily oral micronized progesterone is effective in preventing recurrent spontaneous preterm birth (RSPB) and whether micronized progesterone use increases maternal serum progesterone levels.

DETAILED DESCRIPTION:
To evaluate whether 400 mg daily oral micronized progesterone from 16 to 34 weeks' is effective in preventing recurrent spontaneous preterm birth (RSPB) and whether micronized progesterone use increases maternal serum progesterone levels.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women less than 20 weeks' gestation who had at least one prior spontaneous preterm birth of a liveborn baby between 20 & 0/7 weeks' and 36 & 6/7 weeks' gestation.

Exclusion Criteria:

* multiple gestations, the presence of major fetal anomalies, progesterone use in the current pregnancy (ongoing or past), the presence of a cervical cerclage, and the presence of a placenta previa.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S McKenna, MD, Principal Investigator — Fetal Medicine Foundation/USA
Locations (1):
- Miami Valley HospitaL, Dayton, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Progesterone Group: 400 mg oral micronized progesterone daily at bedtime from 16 to 34 weeks or delivery
- Placebo: Placebo tablets identical to 400 mg micronized progesterone study drug taken daily at bedtime from 16 to 34 weeks or delivery
Period: Overall Study
Arm/Group | Progesterone Group | Placebo
Started | 20 | 16
Completed | 19 | 14
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone Group | Placebo | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 16 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (4.7) | 27.2 (4.9) | 28 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 16 | 36

OUTCOME MEASURES:

1. Primary Outcome: Rate of Recurrent Preterm Birth
Description: Spontaneous preterm birth prior to 37 weeks' gestation. Indicated preterm deliveries (for maternal or fetal reasons) were excluded.
Time Frame: Prior to 37 weeks' gestation
Measure: Number; unit: participants
Arm/Group | Progesterone Group | Placebo
Number analyzed (Participants) | 19 | 14
participants | 5 | 8

2. Secondary Outcome: Secondary Outcomes
Description: Serum progesterone levels
Time Frame: Mean +/- Std Dev gestational age of 25.9/-2.4 weeks in Progesterone group, and 28.4 +/-4.7 weeks in placebo group
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Progesterone Group: oral micronized progesterone: 400 mg oral micronized progesterone nightly from 16 to 34 weeks vs placebo
- Placebo: Identical Placebo tablet: placebo taking nightly from 16 to 34 weeks
Arm/Group | Progesterone Group | Placebo
Number analyzed (Participants) | 15 | 8
pg/mL | 122.6 (61.8) | 90.1 (38.7)

ADVERSE EVENTS:
Time Frame: From trial entry until delivery of the infant, average (+/- std dev) gestational age at randomization was 18.2 +/- 2.7 weeks for placebo group and 16.9 +/- 2.6 weeks for progesterone group; Average gestational age at delivery was 35.9 +/- 3.8 weeks for placebo group, and 37.0 +/- 2.7 weeks for progesterone group. The average duration adverse events were collected was 17.7 weeks for the placebo group, and 20.1 weeks for the progesterone group.
Description: All subjects were queried by an investigator at every prenatal visit regarding adverse events, and the electronic medical record was searched for any occurrences.
Arm/Group | Progesterone Group | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 0/20 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No